CLINICAL TRIAL: NCT00931697
Title: A Phase I Randomised, Double-Blind Study to Investigate the Safety, Tolerability and Pharmacokinetics of AD 452 [(+)-Mefloquine] Compared With Racemic Mefloquine
Brief Title: Study to Investigate the Safety, Tolerability and Pharmacokinetics of AD 452 [(+)-Mefloquine] Compared With Racemic Mefloquine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Treague Ltd (Industry)
Collaborators: Medicines for Malaria Venture (Other)
Responsible Party: Dr Robert Tansley, Treague Ltd
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P-AD452-023
Record Dates: First submitted 2009-06-29; First posted 2009-07-02 (Estimated); Last update posted 2010-08-03 (Estimated); Status verified 2010-07

CONDITIONS: Healthy Subjects
Keywords: Mefloquine; Malaria; (+) Mefloquine; Pharmacokinetics
MeSH Terms: conditions — Malaria | interventions — Mefloquine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- AD 452 (+) mefloquine (Experimental)
  Interventions: Drug: AD 452 (+) mefloquine
- Racemic mefloquine (Active Comparator)
  Interventions: Drug: Racemic Mefloquine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AD 452 (+) mefloquine — Single dose delivered as over-encapsulated tablet at ascending doses
  Arms: AD 452 (+) mefloquine
Drug: Racemic Mefloquine — Single dose delivered as over-encapsulated tablet at ascending dose
  Arms: Racemic mefloquine
Drug: Placebo — Over-encapsulated placebo to maintain blinding
  Arms: Placebo

SUMMARY:
Mefloquine is a quinolinemethanol antimalarial that is effective as therapy and prophylaxis for all species of malaria infecting humans, including multi-drug resistant Plasmodium falciparum. The marketed anti-malaria drug consists of two enantiomers of mefloquine.

Mefloquine's clinical utility has been impaired by its association with neuropsychiatric side effects. The pharmacological basis of mefloquine's side effects is not known but two of the most reported hypotheses relate to its action on (i) the adenosine receptor and (ii) its effect on the cholinesterase enzyme. For both of these mechanisms, there is a significant stereoselective activity of the two enantiomers. In vitro studies show that the (-) isomer is 50-100 fold more potent towards adenosine receptors compared with the (+) isomer. In addition, (-)-mefloquine has considerably more anti-cholinesterase activity. It has therefore been hypothesised that (+)-mefloquine may have a better central nervous system (CNS) safety profile compared with either the racemate or (-)-mefloquine.

This study is a randomized, ascending dose, double-blind, active and placebo-controlled, parallel group study in healthy male and female volunteers designed to investigate this hypothesis and to describe the comparative pharmacokinetics of the racemate and the single enantiomer.

ELIGIBILITY:
Inclusion Criteria:

* A BMI of between 19 and 28
* Negative urine drugs of abuse and breath alcohol test
* Willing to use double barrier contraception for 13 weeks after administration of study drug

Exclusion Criteria:

* Pregnant or lactating females
* Existence of any surgical or medical condition which, in the judgement of the Principal Investigator, might interfere with the absorption and disposition of the drug or with the aim of the study including clinically significant lactose intolerance
* Receipt of prescription medication within 21 days of the first study day or over the counter medication (with the exception of multi-vitamins or paracetamol) within 1 week before the planned dosing date without prior approval
* Definite or suspected personal or family history of adverse drug reaction or hypersensitivity to drugs with a chemical structure similar to AD 452
* Participation in a clinical study within the previous 12 weeks
* A history of sensitivity to antimalarial or related compounds
* Definite or suspected personal or family history of adverse drug reaction or hypersensitivity to drugs with a chemical structure similar to AD 452
* Active depression or a recent history of depression or generalised anxiety disorder
* Any personal history of psychosis or schizophrenia or other major psychiatric disorders or convulsions
* Previous exposure to racemic mefloquine

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2009-06; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
The dose-concentration-effect relationship of AD 452 [(+)-mefloquine] for safety and toleration in comparison with that of racemic mefloquine across a range of potentially therapeutic doses and concentrations. | Following single dose

SECONDARY OUTCOMES:
The comparative pharmacokinetics of AD 452 [(+)mefloquine] and racemic mefloquine | Single dose

CONTACTS AND LOCATIONS:
Overall Officials: Robert Tansley, MBBS, Study Director — Treague Ltd
Locations (1):
- LCG Bioscience, Cambridge, Cambridgeshire, United Kingdom